CLINICAL TRIAL: NCT06273215
Title: Evaluation of the Pharmacokinetics of Microdose Midazolam, Dabigatran, Pitavastatin, Atorvastatin and Rosuvastatin in Diabetic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dongyang Liu, Researcher, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCTC-IIR202217
Record Dates: First submitted 2024-02-12; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Midazolam; Dabigatran; pitavastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-obese T2DM (Experimental)
  Interventions: Drug: The combinations of 10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin were administered to diabetic patients on an empty stomach.
- Obese T2DM (Experimental)
  Interventions: Drug: The combinations of 10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin were administered to diabetic patients on an empty stomach.
- Elderly T2DM (Experimental)
  Interventions: Drug: The combinations of 10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin were administered to diabetic patients on an empty stomach.
- T1DM (Experimental)
  Interventions: Drug: The combinations of 10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin were administered to diabetic patients on an empty stomach.

INTERVENTIONS:
Drug: The combinations of 10 µg midazolam, 375 µg dabigatran etexilate, 10 µg pitavastatin, 50 µg rosuvastatin, and 100 µg atorvastatin were administered to diabetic patients on an empty stomach. — Midazolam, dabigatran etexilate, pitavastatin, rosuvastatin and atorvastatin were provided by the Department of Pharmacy, Peking University Third Hospital, and were dissolved and mixed with normal saline respectively, and the mixing process needed to be fully stirred. Then, according to the concentration of the drug mixed solution, the corresponding volume of mixed solution was given to achieve the dosage of 10 μg midazolam, 375 μg dabigatran etexilate,10 μg pitavastatin, 50 μg rosuvastatin and 100 μg atorvastatin. In order to avoid the food effect, the test drugs were administered on an empty stomach on the administration day in this experiment.

SUMMARY:
1.To explore the functional changes of P-gp, CYP3A4, OATP1B and BCRP in Diabetic patients (including the non-obese T2DM, obese T2DM, elderly T2DM, and T1DM).

ELIGIBILITY:
Inclusion Criteria:

All participants:

1. Patients diagnosed with diabetes prior to trial screening and the duration was more than 1 year, but less than 20 years. Previous diagnostic indicators included, but were not limited to, fasting blood glucose (FBG) ≥7 mmol/L or HbA1c ≥6.5 %.

2. Diabetes with other chronic diseases (e.g., hyperlipidemia or hypertension) but which are well-managed through diet or medication also can be included in study (e.g., systolic blood pressure < 140 mmHg, diastolic blood pressure < 90 mmHg, the low density lipoprotein cholesterol (LDL-C) < 2.6 mmol/L).

3. Signed the Inform Consent Form, fully understood the trial conduction and comply with the requirement of the research.

1. Non-obese Type 2 Diabetes Mellitus (T2DM):

   1. Age between 18-65 (include).
   2. Body mass index (BMI) of 18.5 to 27.9 kg/m2 (include); body weight for male >50 kg, for female >45 kg; the proportion of a specific gender should be no less than one-third.
2. Obese T2DM:

   1. Age between 18-65 (include).
   2. Body mass index (BMI) ≥ 28 kg/m2; body weight for male >50 kg, for female >45 kg; the proportion of a specific gender should be no less than one-third.
3. Elderly T2DM:

   1. Age 75 years or older.
   2. Body mass index (BMI) of 18.5 to 27.9 kg/m2 (include); body weight for male >50 kg, for female >45 kg; the proportion of a specific gender should be no less than one-third.
4. Type 1 Diabetes Mellitus (T1DM):

   1. Patients diagnosed with T1DM prior to trial screening and the duration was more than 1 year, but less than 20 years. Previous diagnostic indicators included, but were not limited to, diabetic patients who need lifelong insulin maintenance therapy or have ketoacidosis tendency or have type 1 diabetes-related autoantibodies (glutamic acid decarboxylase autoantibodies, islet cell antibodies, insulin antibodies, etc.).
   2. Age between 18-65 (include).
   3. Body mass index (BMI) of 18.5 to 27.9 kg/m2 (include); body weight for male >50 kg, for female >45 kg; the proportion of a specific gender should be no less than one-third.

   Exclusion Criteria:

   All participants:

   1. Subjects fasting blood glucose ≥13.3 mmol/L or ≤3.9 mmol/L.

   2. Malignant tumor patient.

   3. History of stroke, chronic seizures, or other neurological disorders.

   4. Combined with serious systemic diseases, such as respiratory, blood, digestive, urinary system diseases.

   5. Participate in any other clinical trial within 3 months prior to the trial.

   6. Blood donation or blood loss ≥400mL or received blood product treatment within 8 weeks prior to the start of the trial.

   7. Family history of clinically significant ECG abnormalities or long QT syndrome.

   8. History of hypersensitive reaction or allergic to study drugs (including Midazolam, Dabigatran etexilate, Pitavastatin, Atorvastatin, and Rosuvastatin).

   9. Patients who could not discontinue the study drugs (including Midazolam, Dabigatran etexilate, Pitavastatin, Atorvastatin, and Rosuvastatin) within 3 days before the trial because of illness.

   10. Take weak/moderate inhibiters or inducers of CYP3A/BCRP/OATP1B/P-gp within 14 days before screening, including but not limited to: clarithromycin, boceprevir, cobicistat, danoprevir, grapefruit juice, indinavir, ketoconazole, telaprevir, paritaprevir, Telithromycin, troleandomycin, voriconazole, nafazodone, Idelalisib, nelfinavir, fluconazole, aprepitant, ciprofloxacin, conivaptan, crizotinib, cyclosporin A, diltiazem, fluvoxamine, imatinib, tofisopam, atazanavir, erythromycin, gemfibrozil, simeprevir, amiodarone, carvedilol, itraconazole, lapatinib, lopinavir, ritonavir, propafenone, quinidine, ranolazine, saquinavir, telaprevir, verapamil, tipranavir, curcumin, Eltrombopag, phenytoin, rifampicin, apalutamide, carbamazepine, St. John's Wort, mitotan, enzalutamide, bosentan, efavirenz, primidone, phenobarbital.

   11. Any condition that may significantly affect the absorption, distribution, metabolism, and excretion of glucose and study drugs, or any condition that may pose a hazard to the subject. Investigators were instructed on the following:

   (1) History of inflammatory bowel disease, gastritis, ulcers, gastrointestinal or rectal bleeding.

   (2) History of major gastrointestinal surgery (e.g., gastrectomy, gastrostomy, or enterectomy).

   (3) Liver function tests (such as ALT, AST) are abnormal and clinically significant, indicating liver disease.

   (4) History or evidence of renal insufficiency manifested; clinically significant creatinine abnormalities or abnormal urine composition (e.g., proteinuria); for non-obese T2DM, obese T2DM, and T1DM, the baseline eGFR < 90 mL/min/1.73m2, and for elderly T2DM, the baseline eGFR < 60 mL/min /1.73m2 (GFR as calculated using the EPI-CKD equation).

   12. Urinary tract obstruction or difficulty emptying during screening.

   13. Subjects who test positive at screening for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HbsAg), and syphilis.

   14. History of drug or alcohol abuse in the 12 months before this study, or evidence of such abuse found on laboratory testing during the screening evaluation.

   15. Smokers are those who smoke more than 10 cigarettes or equivalent per day.

   16. Pregnant or lactating women.

a. Non-obese T2DM:

1. T1DM. 2. BMI≥28 kg/m2.

b. Obese T2DM:

1. T1DM.

c. Elderly T2DM:

1. T1DM. 2. BMI≥28 kg/m2.

d. T1DM:

1. T2DM.
2. BMI≥28 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of study drug | Baseline and within 24 hours after administration
  The plasma concentration of midazolam, dabigatran, pitavastatin, atorvastatin and rosuvastatin before dosing and 1 h, 4 h, 8 h and 24 h.

SECONDARY OUTCOMES:
Concentration of endogenous markers of CYP3A and OATP | Baseline
  The plasma concentration of 4β hydroxycholesterol, cholesterol and coproporphyrin.
Genotype of OATP and BCRP | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China